CLINICAL TRIAL: NCT04251533
Title: A Phase III, Multicenter, Randomized, Double-blind, Placebo-controlled Study to Assess the Efficacy and Safety of Alpelisib (BYL719) in Combination With Nab-paclitaxel in Patients With Advanced Triple Negative Breast Cancer With Either Phosphoinositide-3-kinase Catalytic Subunit Alpha (PIK3CA) Mutation or Phosphatase and Tensin Homolog Protein (PTEN) Loss Without PIK3CA Mutation
Brief Title: Study Assessing the Efficacy and Safety of Alpelisib + Nab-paclitaxel in Subjects With Advanced TNBC Who Carry Either a PIK3CA Mutation or Have PTEN Loss
Acronym: EPIK-B3
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CBYL719H12301; 2019-002637-11 (EudraCT Number)
Record Dates: First submitted 2020-01-30; First posted 2020-02-05 (Actual); Results first posted 2024-07-31 (Actual); Last update posted 2025-11-05 (Actual); Status verified 2025-10

CONDITIONS: Triple Negative Breast Neoplasms
Keywords: Triple Negative Breast Cancer; alpelisib; BYL719; nab-paclitaxel; PIK3CA mutation; PTEN loss
MeSH Terms: conditions — Triple Negative Breast Neoplasms | interventions — Alpelisib; 130-nm albumin-bound paclitaxel; Albumin-Bound Paclitaxel

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Part A: alpelisib + nab-paclitaxel (Experimental): Participants received alpelisib 300 mg orally + nab-paclitaxel 100 mg/m^2 intravenously (IV) on Days 1, 8, and 15 of each 28-day cycle
  Interventions: Drug: alpelisib; Drug: nab-paclitaxel
- Part A: placebo + nab-paclitaxel (Placebo Comparator): Participants received placebo + nab-paclitaxel 100 mg/m^2 IV on Days 1, 8, and 15 of each 28-day cycle.
  Interventions: Drug: placebo; Drug: nab-paclitaxel
- Part B1: alpelisib + nab-paclitaxel (Experimental): Participants received alpelisib 300 mg orally + nab-paclitaxel 100 mg/m^2 IV on Days 1, 8, and 15 of each 28-day cycle.
  Interventions: Drug: alpelisib; Drug: nab-paclitaxel

INTERVENTIONS:
Drug: alpelisib — 300 mg orally, once per day (QD), tablets
  Other Names: BYL719
  Arms: Part A: alpelisib + nab-paclitaxel; Part B1: alpelisib + nab-paclitaxel
Drug: placebo — 300 mg orally, once per day (QD), tablets
  Other Names: alpelisib-matching placebo
  Arms: Part A: placebo + nab-paclitaxel
Drug: nab-paclitaxel — 100 mg/m^2 IV infusion, once per day (QD)
  Other Names: abraxane

SUMMARY:
The purpose of this study was to determine whether treatment with alpelisib in combination with nab-paclitaxel is safe and effective in subjects with advanced triple negative breast cancer (aTNBC) who carry either a PIK3CA mutation (Study Part A) or have PTEN loss (Study Part B1) or PTEN loss without PIK3CA mutation (Study Part B2)

DETAILED DESCRIPTION:
The recruitment of Part A was halted on 11-Nov-2022 due to slow recruitment. Since Part B1 did not meet its primary objective for confirmed overall response rate, the Part B2 was not initiated, and the recruitment was halted for the entire study.

Upon confirming either PIK3CA mutation and/or PTEN loss status, advanced TNBC participants meeting all other eligibility criteria were assigned to either Part A (PIK3CA mutation regardless of PTEN loss) or Part B1 (PTEN loss with PIK3CA unknown or non-mutant).

In Part A, participants were randomized a 1:1 to receive either:

* alpelisib 300 mg daily orally + nab-paclitaxel 100 mg/m^2 intravenously (IV) on Days 1, 8, and 15 of each 28-day cycle or
* placebo + nab-paclitaxel 100 mg/m^2 IV on Days 1, 8, and 15 of each 28-day cycle.

In Part B1, participants received alpelisib 300 mg daily orally + nab-paclitaxel 100 mg/m^2 IV on Days 1, 8, and 15 of each 28-day cycle.

ELIGIBILITY:
Inclusion Criteria:

* Participant has histologically confirmed diagnosis of advanced (loco-regionally recurrent and not amenable to curative therapy), or metastatic (stage IV) TNBC
* Participant has either a measurable disease per RECIST 1.1 criteria or, if no measurable disease is present, then at least one predominantly lytic bone lesion or mixed lytic-blastic bone lesion with identifiable soft tissue component (that can be evaluated by CT/MRI) must be present. Part B1: Participants must have measurable disease
* Participant has adequate tumor tissue to identify the PIK3CA mutation status (either carrying a mutation or without a mutation) and the PTEN loss status; both of which will determine whether the subject can be allocated to Part A - PIK3CA mutation regardless of PTEN status; or to Part B1 - PTEN loss or to Part B2 - PTEN loss without a PIK3CA mutation
* Participant has an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Participant has received no more than one line of therapy for metastatic disease
* Participant has adequate bone marrow and organ function

Exclusion Criteria:

* Participant has received prior treatment with any PI3K, mTOR or AKT inhibitor
* Participant has a known hypersensitivity to alpelisib, nab-paclitaxel or to any of their excipients
* Participant has not recovered from all toxicities related to prior anticancer therapies to NCI CTCAE version 4.03 Grade ≤1; with the exception of alopecia
* Participant has central nervous system (CNS) involvement which was not previously treated and/or was newly detected at screening
* Participant with an established diagnosis of diabetes mellitus type I or uncontrolled type II based on Fasting Plasma Glucose and HbA1c
* Participant has impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of the study drugs (e.g., ulcerative diseases, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome, or small bowel resection) based on investigator discretion
* Participant has a history of acute pancreatitis within 1 year prior to screening or past medical history of chronic pancreatitis
* Participant has currently documented pneumonitis/interstitial lung disease
* Participant has a history of severe cutaneous reactions, such as Steven-Johnson Syndrome (SJS), erythema multiforme (EM),Toxic Epidermal Necrolysis (TEN) or Drug Reaction with Eosinophilia and Systemic Syndrome (DRESS)
* Participant with unresolved osteonecrosis of the jaw

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 137 (Actual)
Dates: Start 2020-06-08 (Actual); Primary Completion 2023-05-31 (Actual); Study Completion 2026-01-13 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (72):
- United States (5):
  - University of California LA, Los Angeles, California
  - Hematology and Oncology Clinic, Baton Rouge, Louisiana
  - Mayo Clinic Rochester, Rochester, Minnesota
  - Park Nicollet Institute, Saint Louis Park, Minnesota
  - SCRI Oncology Partners, Nashville, Tennessee
- Argentina (2):
  - Novartis Investigative Site, Rosario, Santa Fe Province
  - Novartis Investigative Site, CABA
- Australia (2):
  - Novartis Investigative Site, Melbourne, Victoria
  - Novartis Investigative Site, Nedlands, Western Australia
- Austria (2):
  - Novartis Investigative Site, Innsbruck, Tyrol
  - Novartis Investigative Site, Leoben
- Brazil (2):
  - Novartis Investigative Site, Barretos, São Paulo
  - Novartis Investigative Site, São Paulo, São Paulo
- Novartis Investigative Site, Plovdiv, Bulgaria
- China (13):
  - Novartis Investigative Site, Hefei, Anhui
  - Novartis Investigative Site, Shijiazhuang, Hebei
  - Novartis Investigative Site, Changsha, Hunan
  - Novartis Investigative Site, Nanjing, Jiangsu
  - Novartis Investigative Site, Nanchang, Jiangxi
  - Novartis Investigative Site, Changchun, Jilin
  - Novartis Investigative Site, Shengyang, Liaoning
  - Novartis Investigative Site, Shenyang, Liaoning
  - Novartis Investigative Site, Chengdu, Sichuan
  - Novartis Investigative Site, Hangzhou, Zhejiang
  - Novartis Investigative Site, Dalian
  - Novartis Investigative Site, Shanghai
  - Novartis Investigative Site, Tianjin
- Novartis Investigative Site, Bogotá, Colombia
- Novartis Investigative Site, Zagreb, Croatia
- France (4):
  - Novartis Investigative Site, Saint-Cloud, Hauts De Seine
  - Novartis Investigative Site, Angers
  - Novartis Investigative Site, Saint-Herblain
  - Novartis Investigative Site, Villejuif
- Germany (3):
  - Novartis Investigative Site, Dresden, Saxony
  - Novartis Investigative Site, Leipzig, Saxony
  - Novartis Investigative Site, Essen
- Novartis Investigative Site, Budapest, Hungary
- India (4):
  - Novartis Investigative Site, Faridabad, Haryana
  - Novartis Investigative Site, Mumbai, Maharashtra
  - Novartis Investigative Site, Vellore, Tamil Nadu
  - Novartis Investigative Site, Hyderabad, Telangana
- Novartis Investigative Site, Tel Aviv, Israel
- Italy (3):
  - Novartis Investigative Site, Meldola, FC
  - Novartis Investigative Site, Roma, RM
  - Novartis Investigative Site, Napoli
- Malaysia (2):
  - Novartis Investigative Site, Petaling Jaya, Selangor
  - Novartis Investigative Site, Kuala Lumpur
- Novartis Investigative Site, Monterrey, Nuevo León, Mexico
- Novartis Investigative Site, Oslo, Norway
- Novartis Investigative Site, Trujillo, La Libertad, Peru
- Poland (3):
  - Novartis Investigative Site, Gdynia
  - Novartis Investigative Site, Opole
  - Novartis Investigative Site, Poznan
- Russia (4):
  - Novartis Investigative Site, Arkhangelsk
  - Novartis Investigative Site, Chelyabinsk
  - Novartis Investigative Site, Moscow
  - Novartis Investigative Site, Saint Petersburg
- Slovakia (2):
  - Novartis Investigative Site, Bratislava
  - Novartis Investigative Site, Košice
- Novartis Investigative Site, Ljubljana, Slovenia
- South Africa (2):
  - Novartis Investigative Site, Port Elizabeth, Western Cape
  - Novartis Investigative Site, Johannesburg
- Novartis Investigative Site, Seoul, South Korea
- Spain (3):
  - Novartis Investigative Site, Palma, Balearic Islands
  - Novartis Investigative Site, Badajoz, Extremadura
  - Novartis Investigative Site, Alicante
- Novartis Investigative Site, Lausanne, Switzerland
- Novartis Investigative Site, Taipei, Taiwan
- Turkey (Türkiye) (2):
  - Novartis Investigative Site, Istanbul, Fatih
  - Novartis Investigative Site, Istanbul, Kadikoy
- United Kingdom (2):
  - Novartis Investigative Site, Nottingham
  - Novartis Investigative Site, Oxford

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com
URL: https://www.clinicalstudydatarequest.com

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Part A: Alpelisib + Nab-paclitaxel | Part A: Placebo + Nab-paclitaxel | Part B1: Alpelisib + Nab-paclitaxel
Started | 52 | 50 | 35
Completed | 8 | 14 | 4
Not Completed | 44 | 36 | 31
Not completed — Progressive disease | 33 | 29 | 22
Not completed — Death | 5 | 1 | 3
Not completed — Physician Decision | 3 | 2 | 4
Not completed — Participant decision | 1 | 3 | 1
Not completed — Adverse Event | 2 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Part A: Alpelisib + Nab-paclitaxel | Part A: Placebo + Nab-paclitaxel | Part B1: Alpelisib + Nab-paclitaxel | Total
Number analyzed (Participants) | 52 | 50 | 35 | 137
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.8 (9.76) | 59.1 (11.34) | 48.4 (12.21) | 55.5 (11.74)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 52 | 49 | 35 | 136
  Male | 0 | 1 | 0 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 32 | 30 | 23 | 85
  Asian | 17 | 19 | 10 | 46
  Multiple | 1 | 1 | 0 | 2
  Black Or African American | 1 | 0 | 1 | 2
  American Indian or Alaska Native | 0 | 0 | 1 | 1
  Unknown | 1 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival (PFS) Per Investigator Assessment in Study Part A
Description: PFS was defined as time from the date of randomization to the date of the first documented progressive disease (PD) or death due to any cause. PFS was assessed via a local radiology assessment according to RECIST 1.1. PD=At least a 20% increase in the sum of diameter of all measured target lesions, taking as reference the smallest sum of diameter of all target lesions recorded at or after baseline. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm^2. PFS was censored at the date of the last adequate tumor assessment, if no PFS event was observed prior to the analysis cut-off date.
Time Frame: Once all participants have completed at least 6 months of study treatment or have discontinued from study treatment, up to 35 months
Population: Part A: The full analysis set included all participants to whom study treatment was assigned by randomization.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Part A: Alpelisib + Nab-paclitaxel | Part A: Placebo + Nab-paclitaxel
Number analyzed (Participants) | 52 | 50
months | 7.2 [3.71 to 8.57] | 5.6 [3.75 to 12.68]
Statistical Analysis 1: Comparison: Part A: Alpelisib + Nab-paclitaxel vs Part A: Placebo + Nab-paclitaxel; Test type: Superiority; Regression, Cox; Hazard Ratio (HR) = 1.49, 95% CI 2-sided [0.92 to 2.41]

2. Primary Outcome: Overall Response Rate (ORR) Based on Local Radiology Assessments in Participants With Measurable Disease at Baseline in Study Part B1
Description: ORR was defined as the percentage of participants with best overall response (BOR) of confirmed complete response (CR) or confirmed partial response (PR) according to RECIST 1.1. BOR was defined as the best response recorded from the start of the study treatment until progressive disease (PD)/recurrence. CR=Disappearance of all non-nodal target lesions. In addition, any pathological lymph nodes assigned as target lesions must have a reduction in short axis to < 10 mm. PR= At least a 30% decrease in the sum of diameters of all target lesions, taking as reference the baseline sum of diameters; PD= At least a 20% increase in the sum of diameters of all measured target lesions, taking as reference the smallest sum of diameter of all target lesions recorded at or after baseline. In addition, the sum must also demonstrate an absolute increase of at least 5 mm.
Time Frame: Up to 6 months
Population: Part B1: The full analysis set included all participants to whom study treatment was assigned.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Part B1: Alpelisib + Nab-paclitaxel
Number analyzed (Participants) | 35
percentage of participants | 14.3 [4.8 to 30.3]

3. Secondary Outcome: Overall Survival in Study Part A
Description: Overall survival is defined as the time from date of randomization to date of death due to any cause.
Time Frame: Up to 66 months
Reporting Status: Not Posted, anticipated posting 2026-05

4. Secondary Outcome: Overall Response Rate (ORR) With Confirmed Response in Study Part A
Description: ORR with confirmed response was the percentage of participants with best overall response (BOR) of confirmed complete response (CR) or confirmed partial response (PR), as per local review and according to RECIST 1.1. BOR was defined as the best response recorded from the start of the study treatment until progressive disease (PD)/recurrence. CR=Disappearance of all non-nodal target lesions. In addition, any pathological lymph nodes assigned as target lesions must have a reduction in short axis to < 10 mm. PR= At least a 30% decrease in the sum of diameters of all target lesions, taking as reference the baseline sum of diameters; PD= At least a 20% increase in the sum of diameters of all measured target lesions, taking as reference the smallest sum of diameter of all target lesions recorded at or after baseline. In addition, the sum must also demonstrate an absolute increase of at least 5 mm.
Time Frame: as for outcome 1
Population: Part A: The full analysis set included all participants to whom study treatment was assigned by randomization.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Part A: Alpelisib + Nab-paclitaxel | Part A: Placebo + Nab-paclitaxel
Number analyzed (Participants) | 52 | 50
percentage of participants | 40.4 [27.0 to 54.9] | 34.0 [21.2 to 48.8]

5. Secondary Outcome: Clinical Benefit Rate (CBR) With Confirmed Response in Study Part A
Description: Clinical benefit rate (CBR) was defined as the percentage of participants with a best overall response of complete response (CR), or partial response (PR) or an overall lesion response of stable disease (SD), lasting as per local review, for a duration of at least 24 weeks. CR, PR and SD are defined according to RECIST 1.1 based on investigator's assessment. CR: Disappearance of all non-nodal target lesions. In addition, any pathological lymph nodes assigned as target lesions must have a reduction in short axis to < 10 mm PR: At least a 30% decrease in the sum of diameter of all target lesions, taking as reference the baseline sum of diameters. SD: Neither sufficient shrinkage to qualify for PR or CR nor an increase in lesions which would qualify for progressive disease.
Time Frame: as for outcome 1
Population: Part A: The full analysis set included all participants to whom study treatment was assigned by randomization.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Part A: Alpelisib + Nab-paclitaxel | Part A: Placebo + Nab-paclitaxel
Number analyzed (Participants) | 52 | 50
percentage of participants | 50.0 [35.8 to 64.2] | 44.0 [30.0 to 58.7]

6. Secondary Outcome: Clinical Benefit Rate (CBR) With Confirmed Response in Study Part B1
Description: as for outcome 5
Time Frame: Up to 6 months
Population: Part B1: The full analysis set included all participants to whom study treatment was assigned.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Part B1: Alpelisib + Nab-paclitaxel
Number analyzed (Participants) | 35
percentage of participants | 25.7 [12.5 to 43.3]

7. Secondary Outcome: Time to Response (TTR) in Study Part A
Description: Time to response (TTR) was defined as the time from the date of randomization/enrolment to the first documented response of either complete response (CR) or partial response (PR), which must be subsequently confirmed (although date of initial response is used, not date of confirmation). CR and PR were based on tumor response data as per local review and according to RECIST 1.1. CR=Disappearance of all non-nodal target lesions. In addition, any pathological lymph nodes assigned as target lesions must have a reduction in short axis to < 10 mm; PR= At least a 30% decrease in the sum of diameters of all target lesions, taking as reference the baseline sum of diameters.
Time Frame: as for outcome 1
Population: Part A: The full analysis set included all participants to whom study treatment was assigned by randomization.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Part A: Alpelisib + Nab-paclitaxel | Part A: Placebo + Nab-paclitaxel
Number analyzed (Participants) | 52 | 50
months | NA [4.14 to NA] — The median and upper limit of 95% CI were not estimable due to an insufficient number of participants with events. | NA [NA to NA] — The median and lower and upper limit of 95% CI were not estimable due to an insufficient number of participants with events.

8. Secondary Outcome: Time to Response (TTR) in Study Part B1
Description: Time to response (TTR) was defined as the time from the date of randomization/enrolment to the first documented response of either complete response (CR) or partial response (PR), which must be subsequently confirmed (although date of initial response was used, not date of confirmation). CR and PR were based on tumor response data as per local review and according to RECIST 1.1. CR=Disappearance of all non-nodal target lesions. In addition, any pathological lymph nodes assigned as target lesions must have a reduction in short axis to < 10 mm; PR= At least a 30% decrease in the sum of diameters of all target lesions, taking as reference the baseline sum of diameters.
Time Frame: Up to 6 months
Population: Part B1: The full analysis set included all participants to whom study treatment was assigned.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Part B1: Alpelisib + Nab-paclitaxel
Number analyzed (Participants) | 35
months | NA [NA to NA] — The median and lower and upper limit of 95% CI were not estimable due to an insufficient number of participants with events.

9. Secondary Outcome: Duration of Response (DOR) With Confirmed Response in Study Part A
Description: Duration of response (DOR) with confirmed response only applied to participants whose best overall response (BOR) was confirmed complete response (CR) or confirmed partial response (PR) according to RECIST 1.1 based on tumor response data per local review. The start date was the date of first documented response of CR or PR (i.e. the start date of response, not the date when response was confirmed), and the end date was defined as the date of the first documented progressive disease (PD) or death due to underlying cancer. CR=Disappearance of all non-nodal target lesions. In addition, any pathological lymph nodes assigned as target lesions must have a reduction in short axis to < 10 mm; PR= At least a 30% decrease in the sum of diameters of all target lesions, taking as reference the baseline sum of diameters.
Time Frame: as for outcome 1
Population: Part A: The full analysis set included all participants to whom study treatment was assigned by randomization. Results are reported for participants whose best overall response was confirmed complete response (CR) or confirmed partial response (PR).
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Part A: Alpelisib + Nab-paclitaxel | Part A: Placebo + Nab-paclitaxel
Number analyzed (Participants) | 21 | 17
months | 7.39 [5.59 to 9.53] | NA [10.55 to NA] — The median and upper limit of 95% CI were not estimable due to an insufficient number of participants with events.

10. Secondary Outcome: Duration of Response (DOR) With Confirmed Response in Study Part B1
Description: as for outcome 9
Time Frame: Up to approximately 20 months
Population: Part B1: The full analysis set included all participants to whom study treatment was assigned. Results are reported for participants whose best overall response was confirmed complete response (CR) or confirmed partial response (PR).
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Part B1: Alpelisib + Nab-paclitaxel
Number analyzed (Participants) | 5
months | 11.04 [7.46 to NA] — The upper limit of 95% CI was not estimable due to an insufficient number of participants with events.

11. Secondary Outcome: Overall Survival in Study Part B1
Description: Overall survival for Part B1 was defined as the number of participants who were alive at the end of the post-treatment period.
Time Frame: Up to approximately 26 months.
Population: Part B1: All participants to whom study treatment was assigned.
Measure: Count of Participants; unit: Participants
Groups:
- Part B1: Alpelisib + Nab-paclitaxelEdit: Participants received alpelisib 300 mg orally + nab-paclitaxel 100 mg/m^2 IV on Days 1, 8, and 15 of each 28-day cycle.
Arm/Group | Part B1: Alpelisib + Nab-paclitaxelEdit
Number analyzed (Participants) | 35
Participants | 21

12. Secondary Outcome: Progression-free Survival (PFS) Per Investigator Assessment in Study Part B1
Description: PFS was defined as time from the date of enrolment to the date of the first documented progressive disease (PD) or death due to any cause. PFS was assessed via a local radiology assessment according to RECIST 1.1. PD=At least a 20% increase in the sum of diameter of all measured target lesions, taking as reference the smallest sum of diameter of all target lesions recorded at or after baseline. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm^2. PFS was censored at the date of the last adequate tumor assessment, if no PFS event was observed prior to the analysis cut-off date.
Time Frame: Up to 6 months
Population: Part B1: The full analysis set included all participants to whom study treatment was assigned.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Part B1: Alpelisib + Nab-paclitaxel
Number analyzed (Participants) | 35
months | 3.71 [3.15 to 5.88]

13. Secondary Outcome: PFS Based on Local Radiology Assessments Using RECIST 1.1 Criteria for Participants by PIK3CA Mutation Status Measured in Baseline Circulating Tumor Deoxyribonucleic Acid (ctDNA) in Study Part A
Description: PFS in participants with PIK3CA mutation as measured in ctDNA. PFS was defined as time from the date of randomization to the date of the first documented progression or death due to any cause.
Time Frame: as for outcome 1
Population: Part A: The full analysis set included all participants to whom study treatment was assigned by randomization. Results are reported for participants with available data.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Part A: Alpelisib + Nab-paclitaxel | Part A: Placebo + Nab-paclitaxel
Number analyzed (Participants) | 27 | 22
months | 7.5 [3.58 to 9.17] | 3.5 [1.77 to 5.85]

14. Secondary Outcome: Post-Hoc: All Collected Deaths
Description: On-treatment deaths due to any cause were collected from first dose of study medication to 30 days after the last dose of study treatment. Post-treatment survival follow-up deaths were collected from Day 31 after last dose of study medication to the data cut-off date.
Time Frame: On-treatment deaths: Up to approximately 28 months (Part A) or approximately 17 months (Part B1). Post-treatment survival follow-up deaths: Up to approximately 7 additional months (Part A) or approximately 9 additional months (Part B1).
Population: Parts A and B: All participants to whom study treatment was assigned.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Alpelisib + Nab-paclitaxel | Part A: Placebo + Nab-paclitaxel | Part B1: Alpelisib + Nab-paclitaxelEdit
Number analyzed (Participants) | 52 | 50 | 35
Participants
  On-treatment deaths | 6 | 6 | 3
  Post-treatment survival follow-up deaths: number analyzed (Participants) | 46 | 44 | 32
  Post-treatment survival follow-up deaths | 19 | 14 | 11
  All deaths | 25 | 20 | 14

ADVERSE EVENTS:
Time Frame: Adverse events were collected up to approximately 28 months (Part A) or up to approximately 17 months (Part B1). Deaths were collected in the post-treatment survival follow-up from 31 days after last dose of study medication until the data cut-off date, up to approximately 7 additional months (Part A) or approximately 9 additional months (Part B1). These were not considered AEs.
Description: Any sign or symptom that occurred during the conduct of the trial and safety follow-up. Deaths in the post-treatment survival follow-up were not considered adverse events. The total number at risk in the post-treatment survival includes patients that entered the post-treatment survival follow-up period.
Groups:
- Part A: Alpelisib + Nab-paclitaxelEdit: Participants received alpelisib 300 mg orally + nab-paclitaxel 100 mg/m^2 intravenously (IV) on Days 1, 8, and 15 of each 28-day cycle.
- Part A: Placebo + Nab-paclitaxelEdit: Participants received placebo + nab-paclitaxel 100 mg/m^2 IV on Days 1, 8, and 15 of each 28-day cycle.
- Part A: Alpelisib + Nab-paclitaxel (Post-treatment Survival Follow-up); Part A: Placebo + Nab-paclitaxel (Post-treatment Survival Follow-up); Part B1: Alpelisib + Nab-paclitaxel (Post-treatment Survival Follow-up): Deaths collected in the post-treatment survival follow-up period (starting from Day 31 post-treatment). No AEs were collected during this period.
Arm/Group | Part A: Alpelisib + Nab-paclitaxelEdit | Part A: Placebo + Nab-paclitaxelEdit | Part B1: Alpelisib + Nab-paclitaxelEdit | Part A: Alpelisib + Nab-paclitaxel (Post-treatment Survival Follow-up) | Part A: Placebo + Nab-paclitaxel (Post-treatment Survival Follow-up) | Part B1: Alpelisib + Nab-paclitaxel (Post-treatment Survival Follow-up)
All-Cause Mortality (participants affected / at risk) | 6/52 | 6/50 | 3/35 | 19/46 | 14/44 | 11/32
Serious Adverse Events (participants affected / at risk) | 22/52 | 15/50 | 14/35 | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 51/52 | 47/50 | 34/35 | 0/0 | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part A: Alpelisib + Nab-paclitaxelEdit (N=52) | Part A: Placebo + Nab-paclitaxelEdit (N=50) | Part B1: Alpelisib + Nab-paclitaxelEdit (N=35) | Part A: Alpelisib + Nab-paclitaxel (Post-treatment Survival Follow-up) (N=0) | Part A: Placebo + Nab-paclitaxel (Post-treatment Survival Follow-up) (N=0) | Part B1: Alpelisib + Nab-paclitaxel (Post-treatment Survival Follow-up) (N=0)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 1 | 0 | NA | NA | NA
Cataract (Eye disorders) | 1 | 0 | 0 | NA | NA | NA
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1 | NA | NA | NA
Ascites (Gastrointestinal disorders) | 0 | 1 | 0 | NA | NA | NA
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 2 | NA | NA | NA
Haemorrhoids (Gastrointestinal disorders) | 1 | 0 | 1 | NA | NA | NA
Nausea (Gastrointestinal disorders) | 0 | 0 | 1 | NA | NA | NA
Stomatitis (Gastrointestinal disorders) | 3 | 0 | 0 | NA | NA | NA
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1 | NA | NA | NA
Asthenia (General disorders) | 0 | 0 | 1 | NA | NA | NA
Chills (General disorders) | 0 | 1 | 0 | NA | NA | NA
Fatigue (General disorders) | 0 | 1 | 0 | NA | NA | NA
General physical health deterioration (General disorders) | 1 | 0 | 1 | NA | NA | NA
Oedema peripheral (General disorders) | 1 | 0 | 0 | NA | NA | NA
Pain (General disorders) | 1 | 1 | 0 | NA | NA | NA
Peripheral swelling (General disorders) | 0 | 0 | 1 | NA | NA | NA
Pyrexia (General disorders) | 2 | 1 | 0 | NA | NA | NA
Hypertransaminasaemia (Hepatobiliary disorders) | 1 | 0 | 0 | NA | NA | NA
Abscess soft tissue (Infections and infestations) | 0 | 1 | 1 | NA | NA | NA
Anal abscess (Infections and infestations) | 0 | 0 | 1 | NA | NA | NA
Appendicitis perforated (Infections and infestations) | 1 | 0 | 0 | NA | NA | NA
Breast abscess (Infections and infestations) | 0 | 0 | 1 | NA | NA | NA
COVID-19 (Infections and infestations) | 1 | 1 | 1 | NA | NA | NA
Cellulitis (Infections and infestations) | 0 | 1 | 0 | NA | NA | NA
Device related infection (Infections and infestations) | 1 | 0 | 0 | NA | NA | NA
Lower respiratory tract infection (Infections and infestations) | 1 | 1 | 0 | NA | NA | NA
Nasopharyngitis (Infections and infestations) | 0 | 1 | 0 | NA | NA | NA
Osteomyelitis (Infections and infestations) | 0 | 0 | 1 | NA | NA | NA
Pneumonia (Infections and infestations) | 2 | 0 | 1 | NA | NA | NA
Postoperative wound infection (Infections and infestations) | 0 | 1 | 0 | NA | NA | NA
Sepsis (Infections and infestations) | 1 | 0 | 0 | NA | NA | NA
Blood creatinine increased (Investigations) | 1 | 0 | 0 | NA | NA | NA
Lymphocyte count decreased (Investigations) | 0 | 1 | 0 | NA | NA | NA
Weight decreased (Investigations) | 1 | 0 | 0 | NA | NA | NA
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0 | NA | NA | NA
Diabetic metabolic decompensation (Metabolism and nutrition disorders) | 0 | 0 | 1 | NA | NA | NA
Hyperglycaemia (Metabolism and nutrition disorders) | 2 | 0 | 0 | NA | NA | NA
Hypernatraemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | NA | NA | NA
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0 | 1 | NA | NA | NA
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0 | 1 | NA | NA | NA
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 1 | 1 | NA | NA | NA
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | NA | NA | NA
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | NA | NA | NA
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | NA | NA | NA
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | NA | NA | NA
Spinal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | NA | NA | NA
Infected neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1 | NA | NA | NA
Brain oedema (Nervous system disorders) | 0 | 1 | 0 | NA | NA | NA
Haemorrhage intracranial (Nervous system disorders) | 1 | 0 | 0 | NA | NA | NA
Headache (Nervous system disorders) | 0 | 1 | 0 | NA | NA | NA
Bronchial fistula (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | NA | NA | NA
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | NA | NA | NA
Hydrothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | NA | NA | NA
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 4 | 1 | 1 | NA | NA | NA
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | NA | NA | NA
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | NA | NA | NA
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | NA | NA | NA
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | NA | NA | NA
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | NA | NA | NA
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Part A: Alpelisib + Nab-paclitaxelEdit (N=52) | Part A: Placebo + Nab-paclitaxelEdit (N=50) | Part B1: Alpelisib + Nab-paclitaxelEdit (N=35) | Part A: Alpelisib + Nab-paclitaxel (Post-treatment Survival Follow-up) (N=0) | Part A: Placebo + Nab-paclitaxel (Post-treatment Survival Follow-up) (N=0) | Part B1: Alpelisib + Nab-paclitaxel (Post-treatment Survival Follow-up) (N=0)
Anaemia (Blood and lymphatic system disorders) | 25 | 22 | 11 | NA | NA | NA
Leukocytosis (Blood and lymphatic system disorders) | 0 | 0 | 2 | NA | NA | NA
Leukopenia (Blood and lymphatic system disorders) | 10 | 6 | 4 | NA | NA | NA
Lymphopenia (Blood and lymphatic system disorders) | 1 | 3 | 3 | NA | NA | NA
Neutropenia (Blood and lymphatic system disorders) | 10 | 13 | 8 | NA | NA | NA
Tachycardia (Cardiac disorders) | 0 | 1 | 2 | NA | NA | NA
Abdominal pain (Gastrointestinal disorders) | 3 | 2 | 0 | NA | NA | NA
Abdominal pain upper (Gastrointestinal disorders) | 1 | 1 | 2 | NA | NA | NA
Constipation (Gastrointestinal disorders) | 7 | 6 | 7 | NA | NA | NA
Diarrhoea (Gastrointestinal disorders) | 33 | 11 | 21 | NA | NA | NA
Dyspepsia (Gastrointestinal disorders) | 3 | 0 | 5 | NA | NA | NA
Flatulence (Gastrointestinal disorders) | 0 | 0 | 2 | NA | NA | NA
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 1 | 3 | NA | NA | NA
Haemorrhoids (Gastrointestinal disorders) | 1 | 0 | 2 | NA | NA | NA
Nausea (Gastrointestinal disorders) | 20 | 12 | 17 | NA | NA | NA
Stomatitis (Gastrointestinal disorders) | 13 | 2 | 7 | NA | NA | NA
Vomiting (Gastrointestinal disorders) | 13 | 6 | 4 | NA | NA | NA
Asthenia (General disorders) | 9 | 5 | 4 | NA | NA | NA
Fatigue (General disorders) | 12 | 10 | 9 | NA | NA | NA
Malaise (General disorders) | 3 | 0 | 1 | NA | NA | NA
Mucosal inflammation (General disorders) | 5 | 2 | 3 | NA | NA | NA
Oedema peripheral (General disorders) | 4 | 8 | 5 | NA | NA | NA
Peripheral swelling (General disorders) | 3 | 2 | 2 | NA | NA | NA
Pyrexia (General disorders) | 7 | 5 | 4 | NA | NA | NA
Hypersensitivity (Immune system disorders) | 0 | 1 | 2 | NA | NA | NA
COVID-19 (Infections and infestations) | 4 | 11 | 3 | NA | NA | NA
Nasopharyngitis (Infections and infestations) | 0 | 2 | 2 | NA | NA | NA
Paronychia (Infections and infestations) | 0 | 1 | 2 | NA | NA | NA
Upper respiratory tract infection (Infections and infestations) | 5 | 0 | 0 | NA | NA | NA
Urinary tract infection (Infections and infestations) | 4 | 4 | 2 | NA | NA | NA
Alanine aminotransferase increased (Investigations) | 7 | 3 | 4 | NA | NA | NA
Alpha hydroxybutyrate dehydrogenase increased (Investigations) | 0 | 0 | 2 | NA | NA | NA
Aspartate aminotransferase increased (Investigations) | 9 | 8 | 3 | NA | NA | NA
Blood alkaline phosphatase increased (Investigations) | 3 | 3 | 3 | NA | NA | NA
Blood creatine phosphokinase increased (Investigations) | 4 | 1 | 1 | NA | NA | NA
Blood creatinine increased (Investigations) | 6 | 0 | 4 | NA | NA | NA
Blood insulin increased (Investigations) | 1 | 3 | 0 | NA | NA | NA
Blood lactate dehydrogenase increased (Investigations) | 2 | 0 | 4 | NA | NA | NA
Gamma-glutamyltransferase increased (Investigations) | 9 | 9 | 4 | NA | NA | NA
Lipase increased (Investigations) | 3 | 0 | 1 | NA | NA | NA
Lymphocyte count decreased (Investigations) | 2 | 3 | 1 | NA | NA | NA
Neutrophil count decreased (Investigations) | 11 | 12 | 3 | NA | NA | NA
Platelet count decreased (Investigations) | 4 | 3 | 1 | NA | NA | NA
Weight decreased (Investigations) | 24 | 5 | 13 | NA | NA | NA
White blood cell count decreased (Investigations) | 12 | 9 | 3 | NA | NA | NA
Decreased appetite (Metabolism and nutrition disorders) | 13 | 5 | 7 | NA | NA | NA
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0 | 3 | NA | NA | NA
Hyperglycaemia (Metabolism and nutrition disorders) | 38 | 8 | 19 | NA | NA | NA
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 | 1 | 2 | NA | NA | NA
Hyperuricaemia (Metabolism and nutrition disorders) | 1 | 3 | 1 | NA | NA | NA
Hypoalbuminaemia (Metabolism and nutrition disorders) | 2 | 2 | 3 | NA | NA | NA
Hypocalcaemia (Metabolism and nutrition disorders) | 3 | 2 | 3 | NA | NA | NA
Hypokalaemia (Metabolism and nutrition disorders) | 12 | 3 | 5 | NA | NA | NA
Hyponatraemia (Metabolism and nutrition disorders) | 3 | 2 | 3 | NA | NA | NA
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 | 9 | 4 | NA | NA | NA
Back pain (Musculoskeletal and connective tissue disorders) | 6 | 7 | 4 | NA | NA | NA
Muscle spasms (Musculoskeletal and connective tissue disorders) | 3 | 1 | 1 | NA | NA | NA
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 2 | NA | NA | NA
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 2 | 2 | NA | NA | NA
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 3 | 2 | NA | NA | NA
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 6 | 1 | NA | NA | NA
Dizziness (Nervous system disorders) | 3 | 4 | 4 | NA | NA | NA
Dysgeusia (Nervous system disorders) | 2 | 1 | 2 | NA | NA | NA
Headache (Nervous system disorders) | 5 | 4 | 5 | NA | NA | NA
Hypoaesthesia (Nervous system disorders) | 0 | 3 | 1 | NA | NA | NA
Lethargy (Nervous system disorders) | 3 | 2 | 1 | NA | NA | NA
Neuropathy peripheral (Nervous system disorders) | 4 | 6 | 3 | NA | NA | NA
Peripheral sensory neuropathy (Nervous system disorders) | 3 | 3 | 3 | NA | NA | NA
Polyneuropathy (Nervous system disorders) | 1 | 3 | 1 | NA | NA | NA
Taste disorder (Nervous system disorders) | 3 | 0 | 2 | NA | NA | NA
Tremor (Nervous system disorders) | 0 | 1 | 2 | NA | NA | NA
Insomnia (Psychiatric disorders) | 3 | 6 | 2 | NA | NA | NA
Breast pain (Reproductive system and breast disorders) | 2 | 4 | 0 | NA | NA | NA
Cough (Respiratory, thoracic and mediastinal disorders) | 9 | 7 | 5 | NA | NA | NA
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 | 2 | 5 | NA | NA | NA
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 5 | NA | NA | NA
Productive cough (Respiratory, thoracic and mediastinal disorders) | 5 | 1 | 1 | NA | NA | NA
Alopecia (Skin and subcutaneous tissue disorders) | 13 | 14 | 8 | NA | NA | NA
Dry skin (Skin and subcutaneous tissue disorders) | 4 | 1 | 2 | NA | NA | NA
Pruritus (Skin and subcutaneous tissue disorders) | 6 | 5 | 5 | NA | NA | NA
Rash (Skin and subcutaneous tissue disorders) | 13 | 13 | 3 | NA | NA | NA
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 5 | 0 | 2 | NA | NA | NA
Hypertension (Vascular disorders) | 2 | 1 | 2 | NA | NA | NA
Lymphoedema (Vascular disorders) | 2 | 0 | 2 | NA | NA | NA

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2023-03-14): https://cdn.clinicaltrials.gov/large-docs/33/NCT04251533/Prot_000.pdf
  • Statistical Analysis Plan (2023-07-03): https://cdn.clinicaltrials.gov/large-docs/33/NCT04251533/SAP_001.pdf